CLINICAL TRIAL: NCT00231218
Title: the Effectiveness of Echinacea, Propolis and Vitamin C in the Prevention of Respiratory Tract Infections and Gastroenteritis in Preschool Age Children: a Prospective Study
Brief Title: Echinacea, Propolis and Vitamin C for URI Prevention in Preschoolers
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 8348
Record Dates: First submitted 2005-09-30; First posted 2005-10-04 (Estimated); Last update posted 2006-12-14 (Estimated); Status verified 2006-12

CONDITIONS: Common Cold; Gastroenteritis
Keywords: vitamin c; echinacea; propolis; upper respiratory tract infection; common cold; gastroenteritis; dietary supplement; herbal remedy
MeSH Terms: conditions — Common Cold; Gastroenteritis; Respiratory Tract Infections | interventions — Propolis; Ascorbic Acid

INTERVENTIONS:
Drug: dietary supplement--echinacea, propolis, and vitamin c

SUMMARY:
We hypothesize the herbal preparation will enhance the preschoolers' immune response and when taken prophylactically for 12 weeks will decrease episodes of upper respiratory infections and gastroenteritis in the active versus the control group.

DETAILED DESCRIPTION:
This combination of herbs has been studied only once before in preschoolers. In a study of 430 preschoolers reported in Archives of Pediatric and Adolescent Medicine in March of 2004, a similar preparation with a slightly lower dose of Vitamin C decreased upper respiratory infections by 55% (308 to 138). We are repeating this study to see if our results confirm or contradict those of the previous study.

ELIGIBILITY:
Inclusion Criteria:

* Age 3-6

Exclusion Criteria:

* Cystic fibrosis
* Immunodeficiency
* Bronchopulmonary dysplasia
* Anatomic abnormalities of respiratory tract
* Intestinal malabsorption
* Allergy to sunflower seeds

Ages: 3 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 104
Dates: Start 2006-01; Study Completion 2006-03

PRIMARY OUTCOMES:
upper respiratory tract infections

SECONDARY OUTCOMES:
gastroenteritis

CONTACTS AND LOCATIONS:
Overall Officials: michael l macknin, m.d., Study Director — The Cleveland Clinic
Locations (1):
- Cleveland Clinic Foundation, Cleveland, Ohio, United States